CLINICAL TRIAL: NCT03217214
Title: Investigation of a Non-invasive/ Minimally Contact Based Method for Diagnosis of Cardiovascular Disease: Blockage(Stenosis) and Blood Flow
Brief Title: Investigation of Contact Based Method for Diagnosis of Cardiovascular Disease
Acronym: INDICES
Status: Completed | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Nanyang Technological University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/2119
Record Dates: First submitted 2017-07-11; First posted 2017-07-14 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2018-10

CONDITIONS: Carotid Artery Diseases
MeSH Terms: conditions — Carotid Artery Diseases | interventions — Thermography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EP-PT: Existing Procedure EP- Passive Thermography PT (40 patients)
  Passive Thermography (PT): 2 thermoscans of the following parts:
  1. Both carotid artery on left and right of the neck.
  2. Both superficial temporal artery on the left and right of forehead.
  3. Left forearm. No relaxation time will be given between the two tests. Each thermoscanning of region will take 60 seconds. The complete procedure will take 10-15 minutes of time.
  Interventions: Diagnostic Test: Thermography
- EP-ATLIC/ATPC: Existing Procedure EP- Active Thermography ATLIC/ATPC (60 patients)
  Active Thermography (AT): Temperature mapping over both carotid arteries will be done with the application of maximum cooling for 45-60 seconds in pulsed or lock-in manner. Pulsed mode is continuous, lock-in cooling will be intermittent. Maximum cooling time is 45-60 seconds, using a cooling pad/ cold air blower. Continuous thermoscanning will be done from the instance of application of cooling to reaching of a fixed temperature during rewarming. Procedure will be done 2 times per subject on both carotid arteries. Relaxation time between procedures is 10 minutes. A warming pad/ hot air blower will be used after the test to bring the skin temperature to normal. The complete procedure will take 60 min.
  Interventions: Diagnostic Test: Thermography

INTERVENTIONS:
Diagnostic Test: Thermography — Passive thermography for Phase I subjects and Active Thermography for Phase II subjects

SUMMARY:
In the proposed method of sensing the vital health sign related to cardiovascular diseases, thermal heat transfer performance of the skin will be evaluated using a non-contact based Infra-Red temperature sensor. The temperature of the skin is significantly dependent upon the heat source as blood vessels (veins and capillaries) in the vicinity of the skin. However, there are several locations in the human body, where arteries are also at a relatively less depth from the outer skin surface (radial or ulnar arteries at the wrist and carotid artery in the neck). If it is possible to track the flow of blood from the thermal performance of the skin, then it could be useful in predicting various states of the human health related to cardiovascular activities.

Subjects will undergo Existing Procedure EP- Passive Thermography PT for Phase I and Existing Procedure EP- Active Thermography ATLIC/ATPC for Phase II, with Duplex Ultrasound being the existing procedure that is considered as more reliable in clinical practice. Existing Passive Thermography will be used to setup the baseline data for Phase I. The currently under-development temperature mapping method (Active Thermography) that involves application of cooling (either pulsed or lock-in cooling) over the skin will be utilized for Phase II.

DETAILED DESCRIPTION:
HYPOTHESIS AND OBJECTIVES In the proposed method of sensing the vital health sign related to Cardiovascular diseases, thermal heat transfer performance of the skin will be evaluated using a non-contact based Infrared temperature sensor. The temperature of the skin is significantly dependent upon the heat source as blood vessels (veins and capillaries) in the vicinity of the skin. However, there are several locations in the human body, where arteries are also at a relatively less depth from the outer skin surface (radial or ulnar arteries at the wrist and carotid artery in the neck). In any scenario, if it is possible to track the flow of blood from the thermal performance of the skin, then it could be useful in predicting various states of the human health related to cardiovascular activities.

* In the proposed hypothesis, a momentarily higher heat transfer window will be created using localized cooling of a small section of the skin over the superficial blood vessel (minimally contact) and hence, the warming process will be tracked using a non-contact and non-invasive Infrared temperature sensor. With the formation of plaques in the arteries at main aorta, carotid bifurcation or anywhere in the vessel, the flow turns into chaotic turbulent kind or in the case of blockage a very low or no blood flow, which impacts the heat transfer from the blood flow and can be easily detected from the heat transfer over the skin during that momentarily higher heaty transfer window.
* In order to apply this approach to Cardiovascular diseases diagnosis one of the probable method could be scanning temperature change at two locations of the body:

  1. On both carotid artery on left and right of the neck.
  2. On both superficial temporal artery on the left and right of the forehead.
  3. It is expected that skin thermal variation at the forearm will always be in a relation to the blood flow in carotid artery for a healthy person that could be used as a signature marker for an individual to make comparison. Therefore, temperature mapping of the left forearm (upper limb).

This study involves 3 different techniques to be tested on 100 human subjects. Existing procedure to be used will be readily available Duplex Ultrasound that is considered as more reliable in clinical practice. Since the new technology involves temperature mapping, existing potential thermography technique (Passive Thermography) will be used to setup the baseline data. Other than this, currently under-development temperature mapping method (Active Thermography) that involves application of cooling (either pulsed or lock-in cooling) over the skin will be utilized. Accordingly, the whole study is divided into two parts: phase-1 and phase-2 as shown in Figure 2. By the time, the Active Thermography technique will be developed; data collection with the techniques mentioned in phase-1 will be completed.

Phase-1

Existing Technology: Duplex Ultrasound exam will be done on all the subjects to divide them into two groups as healthy and diseased.

Passive Thermography (PT): The study procedures involve taking 2 thermoscans of the following parts:

1. Both carotid artery on left and right of the neck.
2. Both superficial temporal artery on the left and right of the forehead.
3. Left forearm (upper limb).

No relaxation time will be given between any of the two tests. Each thermoscanning of individual regions of measurement (ROM) will take around 60 seconds. The complete procedure will take around 10-15 minutes of time.

Phase-2

Existing Technology: Duplex Ultrasound exam will be done on all the subjects to divide them into two groups as healthy and diseased.

Active Thermography (AT): For this case, temperature mapping over both carotid arteries will be done with the application of maximum cooling (within comfort limit) for 45-60 seconds either in pulsed or lock-in manner. While pulsed mode is the continuous application of cooling, lock-in cooling will be intermittent. The frequency of application of cooling under lock-in cooling method is yet to be decided. However, for both the methods, maximum cooling time will remain fixed as 45-60 seconds. The final cooling method to be used is yet to be decided. Cooling will be done either through a cooling pad or using a cold air blower. The temperature of the cooling fluid in the cooling pad and air for the blower will be maintained in the range of 0oC to 5oC (provisionally), respectively. Due to application of cooling, the localized skin tissue will cool down and start rewarming to attain equilibrium temperature with the ambient as earlier (before application of cooling). A continuous thermoscanning will be done from the instance of application of cooling to the reaching of a fixed temperature (to be decided) during the rewarming. However, the maximum acquisition time after the removal of cooling will be kept fixed to 180 seconds. This procedure will be done 2 times for each subject on both carotid arteries. The relaxation time between every procedure will be 10 minutes. A warming pad or hot air blower will be used after every run of the test so as to quickly bring the skin temperature to normal. Temperature of the hot fluid in the warming pad or warm air through blower will be kept slightly higher than room temperature but less than body core temperature (provisionally in the range of 25oC to 35 oC). The total time for the complete procedure would be around 60 min.

Taking all the standard clinical procedure care, there is no risk of any adverse condition as the whole process of data collection is completely non-invasive and minimally contact (only for phase-2 study).

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 35 - 70
2. Planned for Duplex carotid artery duplex scan
3. Ability to provide informed consent

Exclusion Criteria:

1. Known significant stenosis / disease in subclavian artery
2. Known multiple stenoses or occlusion in cerebral (carotid / vertebral / intracranial ) circulation

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical indication for Duplex Carotid Ultrasound for arterial stenosis detection
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Skin thermal variation | 2 years
  Flow of blood from thermal performance of the skin can be tracked

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof Lim Soo Teik, MBBS, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No